CLINICAL TRIAL: NCT03472781
Title: Demographics and Clinical Characteristics of Paediatric Intraocular Inflammation in Singapore
Status: Completed | Type: Observational
Sponsor: Singapore National Eye Centre (Other Government)
Responsible Party: Principal Investigator, Samanthila Waduthantri, Resident physician, Singapore National Eye Centre
Other Study IDs: R1428/11/2017
Record Dates: First submitted 2017-12-06; First posted 2018-03-21 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Intraocular Inflammation in Children

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with intraocular inflammation: All children diagnosed with intraocular inflammation at Singapore National Eye center from from January 1989 to January 2017.
  Interventions: Other: No intervention. A retrospective case review

INTERVENTIONS:
Other: No intervention. A retrospective case review — No intervention. A retrospective case review on demographics, etiology, clinical features, diagnosis, secondary complications, treatment and outcomes of intraocular inflammation in children aged 16 years and below that presented to uveitis clinic in Singapore National Eye Centre from January 1989 to January 2017.

SUMMARY:
Data on demographics, etiology, clinical features, diagnosis, secondary complications, treatment and outcomes of intraocular inflammation in children aged 16 years and below that presented to uveitis clinic in Singapore National Eye Centre (SNEC) from January 1989 to January 2017, will be retrieved and analyzed from the uveitis database retrospectively.

The results will be compared with other published studies on different study populations.

DETAILED DESCRIPTION:
Data on demographics, etiology, clinical features, secondary complications, treatment and outcomes of intraocular inflammation in children aged 16 years and below that presented to uveitis clinic in Singapore National Eye Centre (SNEC) from January 1989 to January 2017, will be retrieved from the uveitis database retrospectively.

Data on demographics, etiology, clinical features, diagnosis, secondary complications, treatment and outcomes will be analyzed using statistical software.

The results will be compared with other published studies on different study populations.

The results of this study will lead to an improved clinical practice with better treatment selections and an optimised monitoring protocol for follow up care for our paediatric patients with intraocular inflammation. This will lead to better clinical outcomes and prevention of serious sight threatening complications.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 16 years and below
* Clinical diagnosis of intraocular inflammation

Exclusion Criteria:

•Children with ocular conditions other than intraocular inflammation.

Ages: 1 Day to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 16 years and below diagnosed with intraocular inflammation in years and below that presented to uveitis clinic in Singapore National Eye Centre (SNEC) from January 1989 to January 2017
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Demographics and clinical characteristics of pediatric intraocular inflammation | January 1989 to January 2017
  percentage of ethnic distribution, percentage of age distribution, percentage of etiology, percentage of clinical features, percentage of diagnosis, percentage of secondary complications, percentage of treatment, percentage of outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Samanthila Waduthantri, Principal Investigator — Singapore National Eye Center
Locations (1):
- Singapore national eye center, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
There will be no individual identifiable data retrieved from the database. The research data will be stored in a password protected access controlled personal computer in SNEC.